CLINICAL TRIAL: NCT04461249
Title: Comparison Between the Effect of Latanoprost 0.005%, Travoprost 0.004% and Tafluprost 0.0015% on Diurnal Intraocular Pressure Fluctuation in Patients Having Primary Open-angle Glaucoma
Brief Title: Comparison Between Latanoprost , Travoprost and Tafluprost in Reducing IOP Fluctuation in POAG Patients
Status: Completed | Type: Observational
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Ahmed Essam Faseeh, Resident of Ophthalmology, Kasr El Aini Hospital
Other Study IDs: 411993
Record Dates: First submitted 2020-06-27; First posted 2020-07-08 (Actual); Last update posted 2020-07-08 (Actual); Status verified 2020-07

CONDITIONS: Primary Open Angle Glaucoma
Keywords: Prostaglandin analogues
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Latanoprost; Ophthalmic Solutions; Travoprost; tafluprost

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Latanoprost group: Latanoprost 0.005 % eye drops was given once by night for 3 months for newly diagnosed primary open-angle glaucoma patients.
  Interventions: Drug: Latanoprost 0.005% Ophthalmic Solution
- Travoprost group: Travoprost 0.004 % eye drops was given once by night for 3 months for newly diagnosed primary open-angle glaucoma patients.
  Interventions: Drug: Travoprost 0.004% ophthalmic solution
- Tafluprost group: Tafluprost 0.0015 % eye drops was given once by night for 3 months for newly diagnosed primary open-angle glaucoma patients.
  Interventions: Drug: Tafluprost Ophthalmic 0.0015% Ophthalmic Solution

INTERVENTIONS:
Drug: Latanoprost 0.005% Ophthalmic Solution — Latanoprost eye drops was given to newly diagnosed primary open-angle glaucoma patients once by night and intraocular pressure fluctuation was measured using Goldmann applanation tonometer.
  Other Names: Xalatan
  Groups: Latanoprost group
Drug: Travoprost 0.004% ophthalmic solution — Travoprost eye drops was given to newly diagnosed primary open-angle glaucoma patients once by night and intraocular pressure fluctuation was measured using Goldmann applanation tonometer.
  Other Names: Travatan
  Groups: Travoprost group
Drug: Tafluprost Ophthalmic 0.0015% Ophthalmic Solution — Tafluprost eye drops was given to newly diagnosed primary open-angle glaucoma patients once by night and intraocular pressure fluctuation was measured using Goldmann applanation tonometer.
  Other Names: Saflutan
  Groups: Tafluprost group

SUMMARY:
Elevated IOP is a key risk factor for the progression of glaucoma. IOP is subjected to diurnal fluctuation in healthy individuals and higher fluctuation in POAG . So, once-daily antiglaucoma drugs must have consistent efficacy throughout the day. Prostaglandin analogues (PGAs) have become the first-line drops for medical treatment of glaucoma worldwide. In our study, we compare between the efficacy and tolerability of Latanoprost 0.005%, Travoprost 0.004% and Tafluprost 0.0015% on diurnal IOP fluctuation in patients having POAG, IOP fluctuation was assessed before treatment , then 2 weeks and 6 weeks after. A comparable and significant reduction in IOP fluctuation occurred in the 3 groups. Side effects were mild and tolerable.

ELIGIBILITY:
Inclusion Criteria:

* Both genders aged 18 years or more.
* Newly diagnosed POAG cases having :

IOP more than 21 mmHg Open angle on gonioscopy Showing both structural and functional damage (confirmed with OCT and visual field)

Exclusion Criteria:

* Angle closure glaucoma.
* Secondary glaucomas.
* Advanced glaucoma likely to be uncontrolled on monotherapy or needing a low target IOP.
* History of ocular trauma, laser or intraocular surgery.
* Any other ocular disorder including uveitis and cystoid macular edema.
* Known history of allergy or sensitivity to any components of the study medications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed primary open-angle glaucoma patients presented to the Glaucoma outpatient clinic, Kasr El-Aini hospital, Cairo University.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
To Compare Between the Efficacy of Latanoprost 0.005%, Travoprost 0.004% and Tafluprost 0.0015% on Diurnal Intraocular Pressure Fluctuation in Patients Having Primary Open-angle Glaucoma | 3 months from starting the treatment
  Newly diagnosed primary open-angle glaucoma patients received one of the 3 study medications and intraocular pressure fluctuation measured in mmHg by using Goldmann applanation tonometer was compared to the baseline intraocular pressure and to vompare its efficacy to the other 2 drugs

SECONDARY OUTCOMES:
To Compare Between the 3 drugs regarding their tolerability and assess their side effects. | 3 Months from starting the treatment
  All patients were subjected to full Ophthalmological examination before starting the treatment and were assessed in the follow up visits to detect the tolerability of the drugs and detect the occurrence of side effects as dry eyes using shirmer's test, also red eyes, eye lashes Lengthening, periocular pigmentation were evaluated by photography comparing to the baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El-Aini hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] El Hajj Moussa WG, Farhat RG, Nehme JC, Sahyoun MA, Schakal AR, Jalkh AE, Abi Karam MP, Azar GG. Comparison of Efficacy and Ocular Surface Disease Index Score between Bimatoprost, Latanoprost, Travoprost, and Tafluprost in Glaucoma Patients. J Ophthalmol. 2018 Mar 7;2018:1319628. doi: 10.1155/2018/1319628. eCollection 2018. PMID 29707390